CLINICAL TRIAL: NCT00010491
Title: Acupuncture and Moxa: A Randomized Clinical Trial for Chronic Diarrhea in HIV Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01 AT000146-01M; R01AT000146-01 (NIH); R01AT000146-02 (NIH); NCT00009074 (obsolete NCT alias)
Record Dates: First submitted 2001-02-02; First posted 2001-02-05 (Estimated); Last update posted 2008-03-07 (Estimated); Status verified 2008-03

CONDITIONS: HIV Infections
Keywords: Diarrhea; complementary therapies
MeSH Terms: conditions — HIV Infections; Diarrhea | interventions — Acupuncture Therapy; Moxibustion

INTERVENTIONS:
Procedure: Acupuncture
Procedure: Moxibustion

SUMMARY:
The objective of this study is to test alternative treatment strategies to reduce the frequency of chronic diarrhea among HIV positive individuals. 60 percent of patients with HIV disease in the U.S. will have diarrhea at some point in their illness. Although in general many of the opportunistic infections (OI's) associated with HIV have decreased due to new "drug cocktails", many of these drugs, however, have diarrhea as a side effect. In Asian countries, acupuncture (including moxibustion) has been widely used for the treatment of various gastrointestinal (GI) disorders. However, there are no published studies that test treatment protocols using acupuncture or moxibustion on patients with HIV experiencing chronic diarrhea.

DETAILED DESCRIPTION:
The subjects in the study will be 144 men and women with HIV infection who report experiencing 3 or more episodes of diarrhea (non-pathogen related) per 24 hour period for 3 weeks or more. Subjects will be randomized to one of four experimental intervention conditions: Condition 1 subjects receive true acupuncture and true moxibustion; Condition 2 subjects receive true acupuncture and placebo moxibustion; Condition 3, subjects receive true moxibustion and sham acupuncture; Condition 4( Control Group), subjects receive sham acupuncture and placebo moxibustion. Subjects in Conditions 1,2,3,& 4 will attend 20 scheduled sessions over 24 weeks. Week 1 is a baseline session followed by two sessions per week for weeks 2-8 (sessions 2-15), one session per week for weeks 9, 10, 11 and 12 (sessions 16, 17, 18 & 19) and a final follow-up session at week 24. All subjects will complete daily bowel movement and medication data collection diaries for the duration of the study. Measurement of quality of life and level of functioning will be taken pre-intervention (session 1), week 6 (session 10), week 12 (session 19) and week 24 (session 20). All interventions will be implemented by licensed acupuncturists trained in traditional Chinese medicine. This study is designed to assess the efficacy of two alternative medicine treatments for chronic diarrhea associated with HIV in a prospective, randomized, controlled, blinded, parallel groups study under the intent-to-treat principle. True acupuncture, moxibustion, and combination therapy, in which specific meridian points are stimulated according to protocol, will be compared to each other and with the control group, with one-way ANOVA models for pre-treatment minus post-treatment difference scores for diarrhea frequency and stool consistency as the dependent measures and treatment group assignment (Conditions 1 - 4) as the independent variable. Average pretreatment diarrhea frequency and stool consistency scores will be entered as covariates into these models. Sample size determination for the above analysis, based on preliminary data, with 80% power and a two-tailed type I error rate of .05% by the method of Holm (1979) and a 20% attrition factor indicates the need for 36 subjects assigned to each condition to detect a 0.95-standardized difference between the most extreme experimental conditions.

ELIGIBILITY:
Inclusion Criteria:

* HIV seropositive experiencing non-pathogen related diarrhea 3 or more times per 24 hours for a period of 3 weeks or more.
* Able to speak and read English or Spanish

Exclusion Criteria:

* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-09; Study Completion 2003-08

CONTACTS AND LOCATIONS:
Overall Officials: Joyce K. Anastasi, PhD,RN,LAc, Principal Investigator — School of Nursing
Locations (1):
- Columbia University, New York, New York, United States